CLINICAL TRIAL: NCT06569524
Title: A Double-blind, Placebo Randomized，Phase II Study to Evaluate the Efficacy and Safety of TQA2225/AP025 in Adults With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Efficacy and Safety of Recombinant Human FGF21-Fc Fusion Protein for Injection (TQA2225/AP025) in Adult Subjects With Non-alcoholic Steatohepatitis (NASH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA2225-II-01
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQA2225/AP025 or TQA2225/AP025 Placebo 25mg (Experimental): TQA2225/AP025 or TQA2225/AP025 Placebo administered 25mg by subcutaneous (SC) injection weekly for 48 weeks
  Interventions: Drug: TQA2225/AP025 or TQA2225/AP025 Placebo 25mg
- TQA2225/AP025 or TQA2225/AP025 Placebo 50mg (Experimental): TQA2225/AP025 or TQA2225/AP025 Placebo administered 50mg by subcutaneous (SC) injection weekly for 48 weeks
  Interventions: Drug: TQA2225/AP025 or TQA2225/AP025 Placebo 50mg

INTERVENTIONS:
Drug: TQA2225/AP025 or TQA2225/AP025 Placebo 25mg — To evaluate the efficacy and safety of TQA2225/AP025 (25mg) in patients with Non-Alcoholic Steatohepatitis (NASH)
  Arms: TQA2225/AP025 or TQA2225/AP025 Placebo 25mg
Drug: TQA2225/AP025 or TQA2225/AP025 Placebo 50mg — To evaluate the efficacy and safety of TQA2225/AP025 (50mg) in patients with Non-Alcoholic Steatohepatitis (NASH)
  Arms: TQA2225/AP025 or TQA2225/AP025 Placebo 50mg

SUMMARY:
A randomized, double-blind, placebo-controlled Phase II study，to evaluate the efficacy and safety of TQA2225/AP025 in Patients With Non-Alcoholic Steatohepatitis (NASH)

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate in the study and provide written informed consent.
* Male or female aged 18 ≤ age < 75 at the time of signing the informed consent.
* Must have had prior liver biopsy within 180 days of randomization with fibrosis stage 1 to 3 and a NAS of ≥4 with at least a score of 1 in each of the lobular inflammation and ballooning degeneration.
* Confirmation of ≥10% liver fat content on Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF).
* Weight changes≤5% in the 6 weeks prior to randomization.
* No qualitative change in dose for the drugs listed below:

  1. Antidiabetic treatment if glucagon-like peptide-1 receptor agonists (GLP1 receptor agonists) or sodium-glucose co-transporter-2 inhibitors (SGLT2 inhibitors): for at least 3 months
  2. Vitamin E (if at a dose ≥400 IU/day): for at least 6 months
  3. Statins: for at least 3 months
* Females of childbearing potential must practice a consistent and proper use of highly effective method of contraception throughout the study and for 6 month after treatment discontinuation.

Exclusion Criteria:

* Documented causes of chronic liver disease other than NASH
* Type 1 diabetes or uncontrolled Type 2 diabetes defined as:Hemoglobin A1c ≥9% at screening，Fasting blood glucose≥13.9mmol/l
* Uncontrolled hypertension at Screening (values ≥160/100 mm Hg)
* History or presence of cirrhosis
* Subjects with any type of active malignancy or a history of malignancy (except cervical cancer or non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma and papillary thyroid carcinoma) that has been cured for more than 5 years prior to the screening period;
* Unable or unwilling to undergo liver biopsy according to research requirements.
* History of weight loss surgery within 5 years (inclusive) prior to screening
* A major surgery was performed 3 months prior to signing the Informed Consent Form (ICF), or planned during the study period.
* Have experienced any bone trauma, fracture, or bone surgery within ≤ 2 months prior to screening.
* When screening, according to the results of dual energy X-ray absorptiometry (DXA) examination, it meets the criteria for osteoporosis: T≤ -2.5
* Recent history of drug abuse (defined as ≤ 2 years).
* Patient participating in other clinical trials of drugs or medical devices within 3 months prior to screening.
* Abnormal laboratory test values：ALT or AST >5 × ULN；Serum ALP≥2× ULN；eGFR<60mL/min；INR>1.3× ULN；platelets < LLN.
* Pregnant or breastfeeding women.
* Liver transplantation history or planned liver transplantation
* Contraindications for MRI examination
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of 25 or 50mg TQA2225 vs matching placebo on liver biopsy (NASH CRN score) at Week 48 compared with Baseline | After week 48 of TQA2225/AP025 treatment
  1. Proportion with resolution of NASH (ballooning 0, inflammation 0,1) associated with at least 2-point reduction in NAFLD Activity Score (NAS) without worsening of fibrosis stage OR
  2. Proportion with at least a 1-point improvement in fibrosis stage with no worsening of NAS

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to week 48
  Number and percentage of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (53):
- China (53):
  - Lu'an Traditional Chinese Medicine Hospital, Lu'an, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Beijing You 'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xiamen Traditional Chinese Medicine Hospital, Xiamen, Fujian
  - Wuwei Cancer Hospital of Gansu Province, Wuwei, Gansu
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Liuzhou Liutie Central Hospital, Liuchow, Guangxi
  - YuLin Red Cross Hospital, Yulin, Guangxi
  - Qingyuan Hospital Affiliated to Guangzhou Medical University (Qingyuan People's Hospital), Qingyuan, Guangzhou
  - Baoding First Central Hospital, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Sixth People's Hospital, Zhengzhou, Henan
  - Zhengzhou Third People's Hospital, Zhengzhou, Henan
  - Huazhong University of Science Tongji Hospital, Tongji Medical College, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Chifeng Hospital, Chifeng, Inner Mongolia
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi Fifth People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Ganzhou Fifth People's Hospital, Ganzhou, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area Gongli Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Leshan People's Hospital, Leshan, Sichuan
  - Southwest Medical University Affiliated Hospital, Luzhou, Sichuan
  - Meishan People's Hospital, Meishan, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - The First People's Hospital of Zigong City, Zigong, Sichuan
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Puer People's Hospital, Puer, Yunnan
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Rui'an People's Hospital, Hangzhou, Zhejiang
  - Ningbo Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - Yiwu Central Hospital, Yiwu, Zhejiang
  - Zhoushan Hospital, Zhoushan, Zhejiang
  - Zhoukou Central Hospital, Zhoukou, Zhoukou